CLINICAL TRIAL: NCT05339295
Title: Bioequivalence Study of Levomerc (Levofloxacin) 500 mg Tablet With Tavanic (Levofloxacin) 500 mg Tablets
Brief Title: Bioequivalence Study of Levomerc 500 mg Tablets
Acronym: BABE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: Merck Pvt. Ltd, Pakistan (Unknown); Center for bioequivalence studies and clinical reseach (CBSCR), ICCBS, University of Karachi (Unknown)
Responsible Party: Principal Investigator, Dr. Muhammad Raza Shah, Professor, University of Karachi
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CB-007-LEV-2012/Protocol/1.0
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Healthy; Pharmacokintetics
Keywords: Bioequivalence Study; Pakistani Population; healthy volunteers
MeSH Terms: interventions — Levofloxacin; Tablets; Ofloxacin

STUDY DESIGN:
Intervention Model Description: A single center, open Label, Randomized, Two Way Cross over, Two Period, Two Treatment, two Sequence Bioequivalence Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Levomerc (Levofloxacin) tablets 500 mg
  Interventions: Drug: Levofloxacin 500mg
- Reference Group (Active Comparator): Tavanic (Levofloxacin) tablets 500 mg
  Interventions: Drug: Levofloxacin 500mg

INTERVENTIONS:
Drug: Levofloxacin 500mg — A single dose consisting of one tablet of either test drug (Levomerc 500 mg) or reference drug (Tavanic 500mg) administered to each of the subjects in both Period.
  Other Names: Levomerc (Levofloxacin) tablets 500 mg; Tavanic (Levofloxacin) tablets 500 mg

SUMMARY:
An open Label, Randomized, Two Way Cross over, Two Period, Two Treatment, two Sequence Bioequivalence Study of Levomerc tablets (Levofloxacin) 500 mg compared with Tavanic (Levofloxacin) 500 mg Tablet as reference drug in healthy Pakistani subjects under fasting condition.

DETAILED DESCRIPTION:
The study will be conducted on 24 healthy subjects. The study will comprise of two Periods, I and II, each consisting of 36 hours, 12 hours before and 24 hour after the drug administration. All 24 subjects divided in group of 12 each. One group treated with the test (T) and other one with reference (R) drug in Period I and after the wash out period, the same received the alternate treatment in Period II.

blood samples will be collected for up to 24 hours post dose in each period for plasma analysis of Levofloxacin.

ELIGIBILITY:
Inclusion Criteria:

* All subjects should be healthy and free from any epidemic, contagious or measurable disease (e.g. Malaria, Dengue).
* Age range for inclusion will be 18-50 year.
* BMI for all Subjects will be between 18.5-26.9 kg/ m2.
* Non Smokers, who have not smoked in last 3 months.
* Medical history, physical examination and screening tests must fall in normal range, unless the investigator considers the abnormality to be clinically not significant.
* Clinical laboratory test result should be within a normal range.
* Participants (who can read and understand Urdu) should be able to give informed consent, understand and sign the Informed Consent Form.
* Participants should have adequate organ function (i.e., kidney, liver and heart).

Exclusion Criteria:

* Age and/or BMI out of acceptable range.
* Any active allergic disease or a history of any significant allergic disease (e.g. Rhinitis, dermatitis, asthma).
* Known hypersensitivity to Investigational drug(s).
* Abnormal results of blood and urine tests conducted at screening unless the investigator considers an abnormality to be clinically irrelevant.
* Presence or history of cardiac (e.g. Myocardial Infarction, arrythmia), renal (e.g. renal insufficiency) , hepatic (e.g. hepatic impairment) , organ insufficiency, bone marrow disease, hematological abnormality (e.g. leukemia, anemia), photosensitivity, neurological disorders (e.g. Alzheimer's disease) or gastrointestinal disease known to interfere with the drug absorption, distribution, metabolism or elimination (e.g. dysphagia).
* History or presence of any musculo skeletal disease (e.g. Tendonitis).
* Subject donated blood (450ml) within 12 weeks minimum preceding the study.
* Alcoholic or with a history of chronic alcohol intake or consumed alcohol or Gutka in last 3 months.
* Ingestion of OTC drug, within 14 days of drug administration (e.g. aspirin, ibuprofen).
* History of intake of any prescribed medicine (e.g. captopril, sumatriptan) during a period of 30 days, prior to drug administration day of study.
* Ingestion of investigational drug within 30 days, prior to investigational drug administration in the study.
* Ingestion of any known hepatic or renal clearance altering agents (e.g. erythromycin, cimetidine, barbiturates, phenothiazines, etc.) for a period of 30 days, prior to study initiation.
* Subjects with an uncontrolled medical condition (i.e., hypertension, cardiac arrhythmias, CHF) that places the patient at risk by participating in the study.

xiv. Subjects with known HIV, hepatitis B or C infection or autoimmune diseases.

* History of drug exposure which, in the opinion of Investigator, amounts to drug abuse. -
* Participation in other drug studies within three months prior to study initiation.
* Subjects with any physical/mental disability.
* Limited mental capacity to the extent that the subject is unable to provide legal consent and information regarding the side effects or tolerance of the study drug.
* Pregnancy or breast feeding, women of child bearing age who are not using a recognized form of contraception for at least last 30 days or using hormonal contraception, are also excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-07-11 (Actual); Primary Completion 2012-07-20 (Actual); Study Completion 2012-09-20 (Actual)

PRIMARY OUTCOMES:
maximum plasma concentration | up to 24 hours post dose
  maximum drug concentration in plasma after dose
Time to reach maximum plasma concentration | 0 to 24 hours post dose
  Time required for the drug to reach maximum plasma concentration
AUC | 0-2 4hours
  Area under the time versus plasma drug concentration curve

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Muhammad R Shah, PhD, Principal Investigator — CBSCR, ICCBS, University of Karachi; Naghma Hashmi (Co-PI), PhD, Principal Investigator — CBSCR, ICCBS, University of Karachi
Locations (1):
- Center for Bioequivalence Studies and clinical research (CBSCR), ICCBS, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will only be available to other researchers upon reasonable request to PI keeping the participants' confidentiality intact.